CLINICAL TRIAL: NCT05171335
Title: Neoadjuvant Combination Therapy of Lenvima Plus Transcatheter Arterial Chemoembolization (TACE) for Transplant-Eligible Patients With Large Hepatocellular Carcinoma
Brief Title: Neoadjuvant Combination Therapy of Lenvatinib and TACE for Transplant-Eligible Large Hepatocellular Carcinoma Patients
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Maen Abdelrahim, MD, PhD, Pharm.B, Associate Professor of Medicine in Oncology, Houston Methodist Academic Institute, The Methodist Hospital Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00028690
Record Dates: First submitted 2021-12-10; First posted 2021-12-28 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: lenvatinib; Liver Transplantation; Neoadjuvant Therapy; Liver Neoplasms; liver cancer; liver cancer, adult; transplantation; Chemoembolization, Therapeutic
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lenvatinib in Combination with TACE Prior to Liver Transplantation (Experimental): Regimen of six months neoadjuvant lenvatinib in combination with TACE prior to liver transplantation in patients with hepatocellular carcinoma (HCC) beyond Milan Criteria.
  Interventions: Drug: Lenvatinib; Procedure: Transcatheter Arterial Chemoembolization
- Matched Historical Control Patients (Other): Historical controls will be liver transplant recipients matched on age, etiology of liver disease (viral vs. non-viral), listing tumor size, and number of TACE procedures to cases in the intervention group who receive a transplant.
  Interventions: Procedure: Transcatheter Arterial Chemoembolization

INTERVENTIONS:
Drug: Lenvatinib — Participants will receive approximately six, 28-day cycles of lenvatinib (LENVIMA®, Eisai Inc., Woodcliff Lake, NJ). Lenvatinib will be administered at 12 mg orally once daily for patients with a body weight ≥60 kg and at 8 mg orally once daily for patients with a body weight of <60 kg.
  Administration of lenvatinib will occur at least 2 weeks before the first standard of care TACE procedure and study drug treatment will continue for 6 months. Lenvatinib will be held for 7 days before and 7 days after each TACE. Participants can receive up to 3 TACE procedures per protocol depending on their response and transplantation time.
  Other Names: LENVIMA®
  Arms: Lenvatinib in Combination with TACE Prior to Liver Transplantation
Procedure: Transcatheter Arterial Chemoembolization — Traditional standard of care: Transcatheter Arterial Chemoembolization (TACE) treatment for hepatocellular carcinoma. Chemotherapeutic drug-coated particles are inserted via a catheter into an artery that supplies blood to a tumor where the drug works to cut off blood supply to the tumor.
  Other Names: TACE

SUMMARY:
This study will examine the effects of a six-month regimen of neoadjuvant lenvatinib in combination with transcatheter arterial chemoembolization (TACE) prior to liver transplantation in patients with hepatocellular carcinoma (HCC) beyond Milan Criteria. Clinical, outcomes, and exploratory data will be compared to a matched, retrospective cohort.

DETAILED DESCRIPTION:
HCC is the third leading cause of cancer death worldwide with more than 230,000 cases of HCC since 2000 and an estimated 42,000 new cases next year. The purpose of this trial is to examine if combination therapy of lenvatinib (LENVIMA®, Eisai Inc., Woodcliff Lake, NJ) plus transcatheter arterial chemoembolization (TACE) will promote tumor necrosis evidenced by explant pathology in patients with large HCC (>5 cm). TACE blocks blood supply to the tumor and induces tumor necrosis, but this causes hypoxia and subsequent angiogenesis.

In 2015, HCC was the leading diagnosis among liver transplant recipients (27.2%). Transplantation of patients diagnosed with HCC is largely based on tumor size, since this is thought to correlate with posttransplant outcomes. However, emerging evidence shows that tumor stability or response to locoregional therapy (LRT) can be surrogate markers of favorable biology and improved outcomes following transplantation. LRT, including TACE or radiofrequency ablation, that promote tumor stability (defined as no tumor progression in 6 months) serve as bridging therapies to liver transplantation. In tumors that respond to ablation, LRT further augments the success of liver transplantation and reduces the risk of HCC recurrence post-transplant.

Liver transplantation provides the ultimate curative option for patients with HCC with improved overall survival (OS) and recurrence-free survival (RFS) of 85% and 92% at 4 years, respectively, compared to 18.4% without transplantation. To limit disease progression and promote tumor stability while on the transplant waitlist, patients with unresectable HCC typically undergo neoadjuvant treatment. Although the National Comprehensive Cancer Network (NCCN) guidelines recommend the use of neoadjuvant therapy for the management of HCC, no clear-cut guidelines are given regarding the type of LRT or other therapeutic agents. LRT effectively improves 2-yr OS between 20-60% and TACE can achieve complete response in 65.2% of patients. LRT is utilized for preventing tumor growth while on the waitlist and to downstage large tumors to standard Milan Criteria (reduce tumor size to ≤ 5cm). Based on the United Network of Organ Sharing (UNOS) criteria, down-staging of tumors to Milan allows the addition of artificial Model for End-stage Liver Disease (MELD) points to patients while waiting for transplantation to decrease their waiting time. Such additional points afford patients with HCC a timely transplantation since they do not exhibit manifestations of liver failure that drives the MELD score toward transplantation.

Large tumors (>5 cm) commonly require multiple TACE procedures and response failure results in dropout/removal from the transplant waiting list. Despite the partial success of TACE, incomplete tumor necrosis following TACE increases the risk of disease progression and drop-out while waiting for transplantation. Thus, robust neoadjuvant therapies that yield superior tumor necrosis are needed to thwart disease progression and reduce dropout from the transplant waitlist. Additionally, achieving superior tumor necrosis may be accompanied by improved OS and RFS post-transplantation.

Lenvatinib is an inhibitor of the kinase activities of vascular endothelial growth factor (VEGF) receptors VEGFR1 (FLT1), VEGFR2 (KDR), and VEGFR3 (FLT4). Lenvatinib inhibits other kinases that have been implicated in pathogenic angiogenesis, tumor growth, and cancer progression in addition to their normal cellular functions, including fibroblast growth factor (FGF) receptors FGFR1, 2, 3, and 4; platelet derived growth factor receptor alpha (PDGFRα), KIT, and RET. Lenvatinib also exhibited antiproliferative activity in hepatocellular carcinoma cell lines dependent on activated FGFR signaling with a concurrent inhibition of FGF receptor substrate 2α (FRS2α) phosphorylation.

Multitargeted tyrosine kinase inhibitors (TKI) restrict tumor angiogenesis and have been successfully utilized as rescue therapy in patients with HCC following failed TACE. TACE blocks blood supply to the tumor and induces tumor necrosis, but this causes hypoxia and subsequent angiogenesis. The antiangiogenesis mechanisms of TKI/VEGF inhibitors may therefore complement the mechanisms of TACE to provide superior tumor necrosis. Investigations of lenvatinib (Lenvima) demonstrate its mechanism of action as an inhibitor of not only VEGF-driven but also fibroblast growth factor (FGF)-driven proliferation and angiogenesis, resulting in anti-tumor activity across diverse HCC models. In clinical trials of patients with unresectable HCC, the REFLECT study demonstrated non-inferiority in OS and significant improvement in time to progress, overall response rate, and progression-free survival with lenvatinib compared to sorafenib. Altogether, these findings suggest that lenvatinib is potentially a potent and successful therapeutic agent that may synergize with TACE to: i) enhance tumor necrosis while on the wait list, ii) reduce the possibility of patient drop-out while awaiting transplantation, and iii) improve OS and RFS of patients after liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) with histologically or cytologically confirmed HCC beyond Milan Criteria
* Must be treatment naïve and eligible for TACE procedure
* Must be on the liver transplant waiting list and not require any other solid organ transplant
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Patients with hepatitis B virus (HBV) infection (as characterized by positive HBV surface antigen and/or anti-hepatitis B core antibodies (HBcAbs) with detectable HBV DNA (≥10 IU/mL or above the limit of detection per local laboratory) must receive antiviral therapy at least after study enrollment per institutional practice to ensure adequate viral suppression (HBV DNA ≤2000 IU/mL). Patients must be managed for 6 months after the last dose of study treatment. Antiviral therapy will be concurrent with lenvatinib.
* Patients with hepatitis C virus (HCV) infection (as characterized by the presence of detectable HCV RNA or anti-HCV antibody) must be managed per local institutional practice and for 6 months after the last dose of study treatment. Antiviral therapy will be concurrent with lenvatinib.
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner while undergoing active treatment up to 1 week after
* Adequate organ and marrow function, as defined below:

  1. Hemoglobin ≥9 g/dL
  2. Platelet count ≥50,000/μL
  3. Total bilirubin ≤3.0
  4. Albumin ≥2 g/dL
  5. International normalized ratio ≤2
  6. Cardiac ejection fraction ≥45%
* Able to swallow orally administered medication
* Capable of signing informed consent form (ICF) and complying with the study protocol, in the investigator's judgement

Exclusion Criteria:

* Mixed hepatocellular-cholangiocarcinoma or HCC within Milan criteria
* Previously received chemotherapy or immunotherapy for HCC
* Child Pugh assessment score greater than or equal to B8
* Uncontrolled blood pressure (BP; Systolic BP>140 mmHg or diastolic BP >90 mmHg) despite an optimized regimen of antihypertensive medication
* Electrolyte abnormalities that have not been corrected
* Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at Screening
* Bleeding or thrombotic disorders or subjects at risk for severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy
* Participants having > 1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours
* Evidence of portal vein thrombosis that precludes the TACE procedure
* History of another primary malignancy except for the following:

  1. Prostate cancer of pathologic stage less than or equal to T2cN0M0 determined from a prior prostatectomy without biochemical recurrence and who, in the opinion of the investigator, are not deemed to require active intervention, or patients with incidental histologic findings of prostate cancer that has not been treated prior to the study and who do not require specific therapy for prostate cancer beyond surgery and also are considered to be at low risk for recurrence per the investigator
  2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  3. Adequately treated carcinoma in situ without evidence of disease
* Active infection, including tuberculosis or human immunodeficiency virus
* Known intolerance to lenvatinib or any of the excipients
* Females who are breastfeeding or pregnant
* Females of childbearing potential who do not agree to use highly effective contraception during the active treatment phase of the study and for 30 days after the last dose of the study treatment
* Males who do not agree to use highly effective contraception during the active treatment phase of the study and for 30 days after the last dose of the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Percent Tumor Necrosis | At time of transplant surgery
  Percent tumor necrosis measured via pathology of explanted liver at time of transplant

SECONDARY OUTCOMES:
Adverse Event Occurrence | At time of first dose of lenvatinib; 1, 2, 3, 4, 5, 6, 7, 8 months after first dose
  Proportion of adverse events with grade 3 or higher score based on the Common Terminology Criteria for Adverse Events (CTCAE) v.5
Response Rate to Lenvatiib | 3, 6, 9, and 12 months after enrollment
  Response rate (RR) of lenvatinib following TACE by assessing radiologic images (relative to baseline scans) using the modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria
Tumor Staging | 3, 6, 9, and 12 months after enrollment
  Proportion of tumors that are down-staged to standard Milan criteria (tumors < 5cm) based on CT/MRI imaging, relative to baseline CT/MRI imaging of abdomen and pelvis.
Serum Biomarkers | At eligibility screening; within 14 days prior to the administration of the first dose of lenvatinib; at time of administration of first dose of lenvatinib; 1, 2, 3, 4, 5, 6, 7, 8 months after first dose
  Concentration of VEGF, VEGF receptor-2, antiopoietin-2, FGF19, and FGF23 in serum.
Microvessel Density | At time of transplant surgery
  Microvessel density of explanted tumor tissue evidenced by CD31 immunohistochemistry.
Explant Biomarkers | At time of transplant surgery
  Concentration of VEGF, VEGF receptor-2, antiopoietin-2, FGF19, and FGF23 on explant tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Maen Abdelrahim, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsiao P, Hsieh KC, Chen YS, Hsu CC, Lo GH, Li YC, Hsieh PM, Lin HY, Wu TC, Yeh JH, Lin CW. Sorafenib with concurrent multiple-line therapies improves overall survival in advanced stage hepatocellular carcinoma. Medicine (Baltimore). 2019 Jun;98(25):e16074. doi: 10.1097/MD.0000000000016074. PMID 31232945
- [Background] Wu FX, Chen J, Bai T, Zhu SL, Yang TB, Qi LN, Zou L, Li ZH, Ye JZ, Li LQ. The safety and efficacy of transarterial chemoembolization combined with sorafenib and sorafenib mono-therapy in patients with BCLC stage B/C hepatocellular carcinoma. BMC Cancer. 2017 Sep 12;17(1):645. doi: 10.1186/s12885-017-3545-5. PMID 28899349
- [Background] Zhang W, Jin K, Wang F, Zhangyuan G, Yu W, Liu Y, Zhang H, Zhang P, Sun B. Differences in the prognostic value of tumor size on hepatocellular cancer-specific survival stratified by gender in a SEER population-based study. United European Gastroenterol J. 2019 Aug;7(7):933-941. doi: 10.1177/2050640619845602. Epub 2019 Apr 24. PMID 31428418
- [Background] White DL, Thrift AP, Kanwal F, Davila J, El-Serag HB. Incidence of Hepatocellular Carcinoma in All 50 United States, From 2000 Through 2012. Gastroenterology. 2017 Mar;152(4):812-820.e5. doi: 10.1053/j.gastro.2016.11.020. Epub 2016 Nov 23. PMID 27889576
- [Background] Lenvima [Package Insert]. Eisai R&D Management Co., Ltd. http://www.lenvima.com/pdfs/prescribinginformation. pdf. Published 2020. Accessed June 12, 2020.
- [Background] Yang JD, Larson JJ, Watt KD, Allen AM, Wiesner RH, Gores GJ, Roberts LR, Heimbach JA, Leise MD. Hepatocellular Carcinoma Is the Most Common Indication for Liver Transplantation and Placement on the Waitlist in the United States. Clin Gastroenterol Hepatol. 2017 May;15(5):767-775.e3. doi: 10.1016/j.cgh.2016.11.034. Epub 2016 Dec 21. PMID 28013117
- [Background] Daoud A, Teeter L, Ghobrial RM, Graviss EA, Mogawer S, Sholkamy A, El-Shazli M, Gaber AO. Transplantation for Hepatocellular Carcinoma: Is There a Tumor Size Limit? Transplant Proc. 2018 Dec;50(10):3577-3581. doi: 10.1016/j.transproceed.2018.04.038. Epub 2018 Apr 18. PMID 30577241
- [Background] Bharat A, Brown DB, Crippin JS, Gould JE, Lowell JA, Shenoy S, Desai NM, Chapman WC. Pre-liver transplantation locoregional adjuvant therapy for hepatocellular carcinoma as a strategy to improve longterm survival. J Am Coll Surg. 2006 Oct;203(4):411-20. doi: 10.1016/j.jamcollsurg.2006.06.016. Epub 2006 Aug 17. PMID 17000383
- [Background] SEER stats. Liver and intrahepatic bile duct cancer. U.S. Department of Health and Human Services, National Institutes of Health, National Cancer Institute. Cancer Stat Facts Web site. https://seer.cancer.gov/statfacts/html/livibd.html. Published 2019. Accessed December 8, 2019.
- [Background] Mazzaferro V, Regalia E, Doci R, Andreola S, Pulvirenti A, Bozzetti F, Montalto F, Ammatuna M, Morabito A, Gennari L. Liver transplantation for the treatment of small hepatocellular carcinomas in patients with cirrhosis. N Engl J Med. 1996 Mar 14;334(11):693-9. doi: 10.1056/NEJM199603143341104. PMID 8594428
- [Background] Young S, Sanghvi T, Lake JJ, Rubin N, Golzarian J. Predicting post-transarterial chemoembolization outcomes: A comparison of direct and total bilirubin serums levels. Diagn Interv Imaging. 2020 Jun;101(6):355-364. doi: 10.1016/j.diii.2019.12.006. Epub 2020 Jan 13. PMID 31948887
- [Background] Lee S, Kang JH, Kim DY, Ahn SH, Park JY, Kim BK, Kim SU, Han KH. Prognostic factors of sorafenib therapy in hepatocellular carcinoma patients with failure of transarterial chemoembolization. Hepatol Int. 2017 May;11(3):292-299. doi: 10.1007/s12072-017-9792-3. Epub 2017 Mar 21. PMID 28324324
- [Background] Matsuki M, Hoshi T, Yamamoto Y, Ikemori-Kawada M, Minoshima Y, Funahashi Y, Matsui J. Lenvatinib inhibits angiogenesis and tumor fibroblast growth factor signaling pathways in human hepatocellular carcinoma models. Cancer Med. 2018 Jun;7(6):2641-2653. doi: 10.1002/cam4.1517. Epub 2018 May 7. PMID 29733511
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] Victor DW 3rd, Monsour HP Jr, Boktour M, Lunsford K, Balogh J, Graviss EA, Nguyen DT, McFadden R, Divatia MK, Heyne K, Ankoma-Sey V, Egwim C, Galati J, Duchini A, Saharia A, Mobley C, Gaber AO, Ghobrial RM. Outcomes of Liver Transplantation for Hepatocellular Carcinoma Beyond the University of California San Francisco Criteria: A Single-center Experience. Transplantation. 2020 Jan;104(1):113-121. doi: 10.1097/TP.0000000000002835. PMID 31233480
- [Background] Highlights of prescribing information: Lenvima. In:2020.
- [Background] Oligane HC, Xing M, Kim HS. Effect of Bridging Local-Regional Therapy on Recurrence of Hepatocellular Carcinoma and Survival after Orthotopic Liver Transplantation. Radiology. 2017 Mar;282(3):869-879. doi: 10.1148/radiol.2016160288. Epub 2016 Sep 27. PMID 27673508
- [Background] Kudo M. Proposal of Primary Endpoints for TACE Combination Trials with Systemic Therapy: Lessons Learned from 5 Negative Trials and the Positive TACTICS Trial. Liver Cancer. 2018 Sep;7(3):225-234. doi: 10.1159/000492535. Epub 2018 Aug 23. No abstract available. PMID 30319982
- [Background] Lencioni R, Llovet JM. Modified RECIST (mRECIST) assessment for hepatocellular carcinoma. Semin Liver Dis. 2010 Feb;30(1):52-60. doi: 10.1055/s-0030-1247132. Epub 2010 Feb 19. PMID 20175033
- [Background] Hastie T, Tibshirani R, Wainwright M. Statistical Learning with Sparsity: The Lasso and Generalizations. Boca Raton, FL: CRC Press; 2015.